CLINICAL TRIAL: NCT02104531
Title: Shoulder Motion Guided Patient Diagnostic and Treatment Classification
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1403E49122
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Rotator Cuff Shoulder Syndrome and Allied Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shoulder Pain: No intervention. Subjects will have a standard static MRI taken of their shoulder, and also complete a series of shoulder motions using video fluoroscopy.
- Healthy Subjects: No intervention. Subjects will receive a standard shoulder MRI and perform shoulder motions while being measured with video fluoroscopy.

SUMMARY:
The investigators purpose is to determine the ability of a low cost, currently available imaging technique to predict shoulder movement disorders and the location of shoulder disease based on motion analysis of subjects with known shoulder disorders.

DETAILED DESCRIPTION:
Shoulder disorders account for the second largest number of musculoskeletal cases in the United States with a large health care burden. The current standard for diagnosis of shoulder disorders is a clinical exam, visual motion assessment and in some cases, costly magnetic resonance (MR) imaging. However, specific tissue pathologies are not always accurately identified, and often not directly linked to the magnitude of dysfunction. There is a need for categorizing or sub-grouping patients based on the underlying movement dysfunctions with which they present. Video fluoroscopy is a common clinical tool that can improve the accuracy of motion analysis. The investigators are using 2-D fluoroscopy, combined with 3-D MR imaging to measure shoulder motion. From the motion analysis we can predict areas of potential soft tissue disease, and compare these to disease locations from MR imaging. The investigators hypotheses is that our motion based predicted disease locations will be significantly associated with disease locations from MR imaging.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects with normal normal shoulder movement and function will be included, age and gender matched to symptomatic subjects.
* Symptomatic subjects will be included if visual shoulder movement deviates from what might be considered normal; they are experiencing shoulder pain with movement, and clinical examination is consistent with soft tissue cumulative trauma to the soft tissues (rotator cuff disease).
* Clinical MR imaging will be used to confirm rotator cuff disease, subacromial bursitis, and/or bicipital tendinitis.

Exclusion Criteria:

* Age outside the accepted range. Contraindications to radiation exposure (pregnancy or possible pregnancy, other recent substantive radiation exposures (CT scanning, treatments involving radiation). Subjects unable to move through at least 90 degrees of shoulder motion will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with shoulder pain and rotator cuff disease, as well as age and gender matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Rotator cuff tendon predicted disease location | baseline
  Measures will predict presence/absence of rotator cuff disease in each of the supraspinatus, infraspinatus, and subscapularis muscles (rotator cuff).
  Subjects are not followed, there is no intervention. The assessment timeframe is dependent on subjects volunteering for the study and can range from 1 month to 10 years from initial onset of their condition.

SECONDARY OUTCOMES:
Shoulder Motion | baseline
  Shoulder joint motion will be assessed as within normal limits, increased or decreased for both rotational and translational motion of the humerus.
  One cross sectional timepoint assessed, subjects are not followed. Timeframe may be 1 month to 10 years from initial symptom onset.
Shoulder functional status | baseline
  Subjects will complete a functional status questionaire regarding their self-reported shoulder function.
  One cross sectional timepoint assessed, subjects are not followed. Timeframe may be 1 month to 10 years from initial symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Ludewig, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States